CLINICAL TRIAL: NCT04370743
Title: Evaluation of Temperature Detecting (Infrared) Cameras and Non-contact (Infrared) Thermometers (NCITs) for Measuring Body Temperatures
Brief Title: Evaluation of Infrared Cameras and Non-contact Infrared Thermometers for Measuring Body Temperatures
Status: Completed | Type: Observational
Sponsor: Quanzeng Wang (U.S. Federal Agency)
Collaborators: University of Maryland, College Park (Other)
Responsible Party: Sponsor-Investigator, Quanzeng Wang, Biomedical Engineer, Food and Drug Administration (FDA)
Organization: Food and Drug Administration (FDA) (U.S. Federal Agency)
Other Study IDs: FDA RIHSC Protocol #16-011R
Record Dates: First submitted 2020-04-25; First posted 2020-05-01 (Actual); Last update posted 2020-05-01 (Actual); Status verified 2020-04

CONDITIONS: Fever
MeSH Terms: conditions — Fever

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

GROUPS / COHORTS (1):
- Group 1
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention

SUMMARY:
Fever is one of the key symptoms exhibited by contagious patients infected with the Ebola and other viruses. Thermographs and non-contact infrared thermometers (NCITs) are commonly used as early detection tools for screening and isolating sick individuals in healthcare settings and transit centers such as airports. The objective of this clinical study is to evaluate the temperature measurement accuracy of thermographs and NCITs. The study will be accomplished by establishing a protocol based on best practices for screening published in the IEC 80601-2-59:2008 Medical electrical equipment -- Part 2-59: Particular requirements for basic safety and essential performance of screening thermographs for human febrile temperature screening standard, performing initial measurements in patients to optimize clinical procedures, then performing quantitative clinical measurements in febrile and afebrile human subjects to compare thermographs - used in accordance with recognized best practices for measurement - with NCITs for fever screening. Since thermographs and NCITs represent the only currently viable mass screening approaches for infectious disease pandemics, like the recent Ebola virus disease (EVD) outbreak in West Africa, the study will evaluate these thermal modalities as medical countermeasures for fever-related pandemics and therefore improve response to these diseases.

ELIGIBILITY:
Inclusion Criteria:

* Any human subject above the age of 18 that can sit for about 40 minutes with permitted breaks as needed and follow the study instructions can be included.

Exclusion Criteria:

* Human subjects should be free of recent (1 week prior) or current disease affecting the ICR and forehead skin. They should not use topical cosmetics, creams or medications on the face on the day of participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Human subject above the age of 18
Sampling Method: Non-Probability Sample
Enrollment: 1125 (Actual)
Dates: Start 2016-11-30 (Actual); Primary Completion 2017-04-28 (Actual); Study Completion 2018-04-25 (Actual)

PRIMARY OUTCOMES:
Evaluating accuracy of infrared cameras and thermometers for skin temperature measurement | Through study completion, about 2 year
  The temperatures of each participant were measured with two infrared (IR) cameras and multiple IR thermometers at different locations on facial skin. The measured temperatures were compared with oral temperature to evaluate the accuracy of IR cameras and IR thermometers.